CLINICAL TRIAL: NCT07292948
Title: The Effect of a Pelvic Floor Training Program on Perineal Trauma During Birth: A Patient-Preference Controlled Clinical Trial
Brief Title: Pelvic Floor Training Program and Perineal Trauma During Vaginal Birth
Acronym: PFTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Incebıyik (Other)
Responsible Party: Sponsor-Investigator, Mehmet Incebıyik, Assistant Professor of Obstetrics and Gynecology, Harran University
Organization: Harran University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HU-PFTP-PERINEAL-TRAUMA-2025
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Perineal Trauma; Pelvic Floor Dysfunction; Labor Complications; Pelvic Floor Muscle Training
Keywords: Pelvic Floor Muscle Training; Perineal Trauma; Obstetric Anal Sphincter Injury; Vaginal Birth; Second Stage of Labor; Postpartum Urinary Incontinence; Antenatal Exercise Program
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two parallel groups based on patient preference: a pelvic floor training group and a standard care control group. Both groups were followed concurrently throughout the study period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors who evaluated perineal trauma and neonatal outcomes were blinded to the participants' group assignments. All other study personnel and participants were aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Training Program (Experimental): Participants in this arm received a structured antenatal pelvic floor muscle training program. The program included twice-weekly supervised PFMT sessions and a daily home-exercise routine from 20 to 34 weeks of gestation. Exercises consisted of sets of maximal voluntary pelvic floor contractions following a standardized protocol. Adherence was monitored through session attendance and weekly follow-up.
  Interventions: Behavioral: Pelvic Floor Muscle Training Program
- Standard Antenatal Care (No Intervention): Participants in this arm received routine antenatal care with no structured pelvic floor muscle training program. They were followed throughout pregnancy and delivery according to standard clinical practice.

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training Program — A structured antenatal pelvic floor muscle training program consisting of twice-weekly supervised sessions and a daily home-exercise routine from 20 to 34 weeks of gestation. Sessions included repeated maximal voluntary pelvic floor contractions following a standardized protocol with progressive intensity. Adherence was monitored through attendance logs and weekly follow-up.
  Other Names: Pelvic Floor Training
  Arms: Pelvic Floor Training Program

SUMMARY:
This study aims to determine whether a structured pelvic floor muscle training program during pregnancy can reduce perineal trauma during vaginal birth. Nulliparous pregnant women at 28 weeks of gestation or later were invited to participate. Women who chose to join the training program performed supervised pelvic floor exercises twice weekly and daily home exercises. Women who declined the program received standard antenatal care.

The study compared rates of severe perineal tears (third- or fourth-degree lacerations), episiotomy, the duration of the second stage of labor, postpartum urinary incontinence, and neonatal outcomes between the two groups. The goal of the study is to evaluate whether pelvic floor training can improve maternal and neonatal birth outcomes.

DETAILED DESCRIPTION:
This prospective, patient-preference controlled clinical trial was conducted to evaluate whether a structured antenatal pelvic floor muscle training (PFMT) program can reduce perineal trauma and improve maternal birth outcomes. Low-risk nulliparous pregnant women at 28 weeks of gestation or later were invited to participate. Women who chose to participate in the training program formed the intervention group, while those who declined received standard antenatal care and served as controls.

The intervention consisted of supervised PFMT sessions twice weekly, combined with a daily home-exercise program. Exercises followed a standardized protocol focusing on repeated maximal voluntary pelvic floor contractions with progressive increases in intensity. Adherence was monitored through attendance records and weekly follow-up.

The study assessed severe perineal trauma (third- or fourth-degree tears) as the primary outcome. Secondary outcomes included episiotomy rate, duration of the second stage of labor, postpartum urinary incontinence, and neonatal outcomes. All participants provided written informed consent, and the study was approved by the institutional ethics committee. The findings aim to inform whether structured PFMT should be incorporated into routine antenatal care to support maternal pelvic floor health and improve labor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous pregnant women aged 18 to 36 years

Singleton pregnancy

Gestational age of 28 weeks or greater at enrollment

Low-risk pregnancy without known obstetric complications

Planning a vaginal delivery

Able and willing to participate in supervised exercise sessions

Exclusion Criteria:

* Multiple gestation

Placenta previa or other contraindications to vaginal birth

Preeclampsia or gestational hypertension

Diabetes requiring medication

History of pelvic floor or urogenital surgery

Neurological disorders affecting continence or pelvic floor function

Inability to attend regular training sessions

Refusal to provide informed consent

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Severe Perineal Trauma (Grade 3-4) | At delivery
  Severe perineal trauma is defined as third- or fourth-degree obstetric anal sphincter injuries (OASIS). Diagnosis is made by the attending clinician immediately after delivery using standard perineal examination and classification procedures.

CONTACTS AND LOCATIONS:
Overall Officials: MEHMET İNCEBIYIK, MD, Study Director — Harran University
Locations (1):
- Harran University Research and Application Hospital, Şanliurfa, HALİLİYE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains identifiable maternal and neonatal information that cannot be publicly released under institutional ethics regulations and national data protection laws. Summary data may be provided upon reasonable request.